CLINICAL TRIAL: NCT00911729
Title: Content Validation of the EORTC QLQ-C30 Version 3.0, and NIH Quality of Life and Symptoms Questionnaire for Pheochromocytoma and Paraganglioma
Brief Title: Content Validation of Quality of Life and Symptom Questionnaires for Pheochromocytoma and Paraganglioma
Status: Terminated | Type: Observational
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Meredith Frank-Molnia, Molecular Insight Pharmaceuticals, Inc
Other Study IDs: A1970
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: paraganglioma; pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this qualitative study is to evaluate the clarity and comprehensiveness of two disease-specific questionnaires, and to evaluate how effective these questionnaires are at assessing the quality of life and symptoms of patients with pheochromocytoma or paraganglioma.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and be willing to comply with protocol requirements
* Participant is aged ≥ 18
* Have a documented (medical record) diagnosis of either pheochromocytoma or paraganglioma with active symptoms or within 60 days of curative therapy

Exclusion Criteria:

Patient is currently asymptomatic from pheochromocytoma/paraganglioma diagnosis or duration > 60 days from curative therapy

* Participant has a clinically significant disorder, including alcohol or drug abuse, which may interfere with study participation or which may affect the outcome of the study as judged by the investigator.
* Participant has a mental disability or significant mental illness, legal incapacity or limited legal capacity or any other lack of fitness, in the investigator's opinion, to preclude the subject's participation in or ability to complete the study.
* Participant is currently too unwell to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a documented (medical record) diagnosis of either pheochromocytoma or paraganglioma with active symptoms or who are within 60 days of curative therapy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2009-04

PRIMARY OUTCOMES:
The main objective of this study is to evaluate content validity of the NIH Quality of Life and Symptoms Questionnaire for Pheochromocytoma and Paraganglioma and EORTC-QLQ-C30 in patients with pheochromocytoma or paraganglioma. | Single Visit

CONTACTS AND LOCATIONS:
Overall Officials: Emuella M Flood, BS, Principal Investigator — Oxford Outcomes
Locations (1):
- Oxford Outcomes- Nationwide Recruitment within the US, Bethesda, Maryland, United States